CLINICAL TRIAL: NCT05396859
Title: A Phase I Study of Entrectinib in Combination With ASTX727 (35 mg Decitabine and 100 mg Cedazuridine) in Patients With Relapsed/Refractory TP53 Mutated Acute Myeloid Leukemia (AML)
Brief Title: Entrectinib in Combination With ASTX727 for the Treatment of Relapsed/Refractory TP53 Mutated Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Genentech, Inc. (Industry); Taiho Oncology, Inc. (Industry)
Responsible Party: Principal Investigator, Ronan Swords, M.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00023205; NCI-2022-02156 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00023205 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-04-20; First posted 2022-05-31 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; entrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ASTX727, entrectinib) (Experimental): Patients receive entrectinib PO QD on days 1-28 and ASTX727 PO QD on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Entrectinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inqovi
Drug: Entrectinib — Given PO
  Other Names: Rozlytrek; RXDX 101; RXDX-101; RXDX101
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of entrectinib when given with ASTX727 in treating patients with acute myeloid leukemia (AML) that has come back (relapsed) or that does not respond to treatment (refractory) and has a genetic change (mutation) in the TP53 gene. ASTX727 is a combination of cedazuridine and decitabine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Entrectinib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals cancer cells to multiply. This helps to stop or slow the spread of cancer cells. Giving ASTX727 and entrectinib together may kill more tumor cells in patients with AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of decitabine and cedazuridine (ASTX727) combined with entrectinib in relapsed/refractory (R/R) AML patients with TP53 mutations.

SECONDARY OBJECTIVE:

I. To assess overall safety and preliminary anti-AML activity of combined ASTX727 and entrectinib regimen.

EXPLORATORY OBJECTIVE:

I. To assess the potential pharmacodynamic changes observed with treatment consisting of entrectinib alone and in combination with decitabine.

OUTLINE: This is a dose-escalation study of entrectinib.

Patients receive entrectinib orally (PO) once daily (QD) on days 1-28 and ASTX727 PO QD on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and willing to sign an informed consent document.
* Participants aged 18 years or older.
* Morphologically documented AML in patients with relapsed/refractory disease, defined as having >= 20% blasts in bone marrow or peripheral blood.
* Documented TP53 mutation as seen on standard diagnostics in AML.
* Aspartate aminotransferase (AST) < 3 × upper limit of normal (ULN).
* Alanine aminotransferase (ALT) < 3 × ULN.
* Total bilirubin < 1.5 × ULN (except for patients with known Gilbert's syndrome).
* Adequate renal function as defined by calculated creatinine clearance (according to the Cockcroft-Gault equation) > 40 mL/min OR serum creatinine < 1.5 × ULN.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2.
* Must be able to take oral medication.
* Individuals of childbearing potential (IOCBP) must agree to use highly-effective method(s) of contraception during the study and six months after the last dose of study drugs. IOCBP must have a negative pregnancy test prior to study enrollment.
* Sperm producing individuals must agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of study drugs.
* Participants must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of their cancer.

Exclusion Criteria:

* Isolated myeloid sarcoma (patients must have blood or marrow involvement with AML to enter the study).
* Acute promyelocytic leukemia (M3).
* Active central nervous system (CNS) involvement by AML.
* Clinical signs/symptoms of leukostasis which has failed urgent therapy of at least 3 days duration, which may have included hydroxyurea or leukapheresis.
* Known active human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C infection.
* Disseminated intravascular coagulopathy with active bleeding or signs of thrombosis.
* Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent or who have agent-related toxicity that has not resolved to grade 1 or less. If the half-life of an investigational agent is unknown, patients must wait 1 week after discontinuing it before receiving the first dose of study treatment. An investigational agent is one for which there is no approved indication by the United States (US) Food and Drug Administration (FDA).
* Prior entrectinib for other malignancies (prior decitabine therapy will not be excluded).
* Patients with psychological, familial, social, or geographic factors that otherwise preclude them from giving informed consent, following the protocol, or potentially hamper compliance with study treatment and follow-up.
* Patients who are otherwise felt unable to comply with the protocol, in the opinion of the investigator.
* Any other significant medical condition, including psychiatric illness or laboratory abnormality, that would preclude the patient participating in the trial or would confound the interpretation of the results of the trial.
* Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic (New York Heart Association [NYHA] class III or IV) congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction at presentation of AML, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
* Patients with uncontrolled infection shall not be enrolled until infection is treated and controlled.
* Participants with prior documented history of malabsorption syndrome (e.g., short gut syndrome) that might limit the bioavailability of study medications will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | From first dose of study drug (day 1 of cycle 0) to end of cycle 1 (each cycle = 28 days)
  Toxicities will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version [v] 5.0).

SECONDARY OUTCOMES:
Incidence of treatment-related grade >= 3 adverse events | From first dose of study drug (day 1 of cycle 0) up to 30 days post end of therapy (each cycle = 28 days)
  Treatment-related grade >= 3 adverse events will be tallied and summarized for the entire safety analysis set and within subgroups defined by each participant's assigned entrectinib dose level. AE tabulations will be constructed at both the participant-level and the event-level, with each toxicity summarized by grade (i.e., severity), duration, and system organ class. AE incidence will be reported using frequency counts and percentages with 95% exact binomial confidence intervals (CIs).
Composite complete remission (CCR) rate | From first dose of study drug up to 2 weeks after last dose of study drug, start of new cancer therapy, or transplant, end of study follow up, death (whichever is first), assessed up to 6 months
  cCR is defined as the proportion of participants who attain a best response of Complete Remission with incomplete blood count recovery (CRi), Complete Remission (CR), or Complete Remission with Minimal Residual Disease (CRMRD) per 2017 European LeukemiaNet (ELN). Each response endpoint will be computed for both the safety analysis set and the efficacy analysis set, with a fraction's numerator equaling the number of participants achieving the requisite degree of response and the denominator comprising the number of participants in the respective analysis set.
Overall response rate (ORR) | From first dose of study drug up to 2 weeks after last dose of study drug, start of new cancer therapy, or transplant (whichever is first), assessed up to 6 months
  Each response endpoint will be computed for both the safety analysis set and the efficacy analysis set, with a fraction's numerator equaling the number of participants achieving the requisite degree of response and the denominator comprising the number of participants in the respective analysis set.
Clinical benefit rate (CBR) | From first dose of study drug up to 2 weeks after last dose of study drug, start of new cancer therapy, or transplant (whichever is first), assessed up to 6 months
  Each response endpoint will be computed for both the safety analysis set and the efficacy analysis set, with a fraction's numerator equaling the number of participants achieving the requisite degree of response and the denominator comprising the number of participants in the respective analysis set.
Proportion transplanted | From first dose of study drug up to end of follow-up or death, assessed up to 6 months
  The proportion of participants in the safety analysis set who transition to stem cell transplantation will be computed and reported as a percentage with a 95% exact CI.
Duration of response (DOR) | From first dose of study drug up to end of follow-up, loss of partial response (PR), progression or death (whichever is first), assessed up to 6 months
  Will be estimated by the Kaplan-Meier method and reported with the median and rates at various landmark times (e.g., 3 months, 6 months, 1 year), each accompanied with a 95% complementary log-log CI.
Event free survival (EFS) | From first dose of study drug up to end of follow-up, relapse, progression, start of new cancer therapy, study drug discontinuation due to toxicity or death (whichever is first), assessed up to 6 months
  Will be estimated by the Kaplan-Meier method and reported with the median and rates at various landmark times (e.g., 3 months, 6 months, 1 year), each accompanied with a 95% complementary log-log CI.
Overall survival (OS) | From first dose of study drug up to end of follow-up or death, assessed up to 6 months
  Will be estimated by the Kaplan-Meier method and reported with the median and rates at various landmark times (e.g., 3 months, 6 months, 1 year), each accompanied with a 95% complementary log-log CI.

OTHER OUTCOMES:
Genomic analysis | Pre-dose Cycle 0; At Cycle 1 day 1; Cycle 1, Day 8; Cycle 1, Day 28 (each cycle = 28 days)
  Expression or intensity changes will be modeled with a paired t-test, linear mixed effects model, or marginal model using a generalized estimating equation.
Total NTRK protein levels | Pre-dose Cycle 0; At Cycle 1 day 1; Cycle 1, Day 8; Cycle 1, Day 28 (each cycle = 28 days)
  Expression or intensity changes will be modeled with a paired t-test, linear mixed effects model, or marginal model using a generalized estimating equation.
NTRK phosphorylation levels | Pre-dose Cycle 0; At Cycle 1 day 1; Cycle 1, Day 8; Cycle 1, Day 28 (each cycle = 28 days)
  Expression or intensity changes will be modeled with a paired t-test, linear mixed effects model, or marginal model using a generalized estimating equation.
RUNX1 protein levels | Pre-dose Cycle 0; At Cycle 1 day 1; Cycle 1, Day 8; Cycle 1, Day 28 (each cycle = 28 days)
  Expression or intensity changes will be modeled with a paired t-test, linear mixed effects model, or marginal model using a generalized estimating equation.
ERK1/2 phosphorylation levels | Pre-dose Cycle 0; At Cycle 1 day 1; Cycle 1, Day 8; Cycle 1, Day 28 (each cycle = 28 days)
  Expression or intensity changes will be modeled with a paired t-test, linear mixed effects model, or marginal model using a generalized estimating equation.
NTRK gene expression | Pre-dose Cycle 0; At Cycle 1 day 1; Cycle 1, Day 8; Cycle 1, Day 28 (each cycle = 28 days)
  Expression or intensity changes will be modeled with a paired t-test, linear mixed effects model, or marginal model using a generalized estimating equation.
RUNX1 gene expression | Pre-dose Cycle 0; At Cycle 1 day 1; Cycle 1, Day 8; Cycle 1, Day 28 (each cycle = 28 days)
  Expression or intensity changes will be modeled with a paired t-test, linear mixed effects model, or marginal model using a generalized estimating equation.

CONTACTS AND LOCATIONS:
Overall Officials: Ronan T Swords, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States